CLINICAL TRIAL: NCT04359160
Title: Comparison of Follow-up by Mobile Application or Paper Questionnaire of Patients Undergoing Rotator Cuff Surgery: Monocentric, Prospective, Randomized Study
Brief Title: Comparison of Follow-up by Mobile App or Paper Questionnaire of Patients Undergoing Rotator Cuff Surgery
Acronym: OFUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L'Institut de Recherche en Chirurgie Orthopédique et Sportive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020 0016 J
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Rotator Cuff Injuries
Keywords: Mobile App; Rotator Cuff; Outpatient surgery; Follow-up
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile-app follow-up (Experimental): The mobile app follow-up group will receive an email, to connect into a secure website. They will answer to periodical questions about their condition. They will have a medical appointment at 6 weeks postoperative and 12 weeks postoperative. All of this information is submitted via the mobile application (Orthense, Digikare Inc. Blagnac, France).The surgeon will have an access to the answer of the patient in real time, and if the patient didn't answer.
  Interventions: Device: Orthense, Orthense, Digikare Inc. Blagnac, France
- Conventional follow-up (Active Comparator): Patients in the conventional, questionnaire follow-up group will have the same periodical questions but on paper. They will have to stick personally with the schedule without any reminders. They will have a medical appointment at 6 weeks postoperative and 12 weeks postoperative where they have to bring the questionnaire.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Device: Orthense, Orthense, Digikare Inc. Blagnac, France — Mobile-app follow-up care, with questions and score
  Arms: Mobile-app follow-up
Other: Questionnaire — Paper questionnaire follow-up, with questions and score
  Arms: Conventional follow-up

SUMMARY:
This study evaluate if in an outpatient rotator cuff surgery, can the use of mobile app compared to conventional paper questionnaire improve follow-up care in the first 90-days following surgery.

DETAILED DESCRIPTION:
Rotator cuff surgery is a painful arthroscopic surgery. In outpatient surgery, the surgeons have to increase the security and surveillance after the surgery to reassure the patient and avoid complications.

Most patients receiving ambulatory rotator cuff surgery have high pain score, and management and aspects of the rehabilitation can be challenging. However, regular follow-up is still considered important in the early post-operative phase. In between the conventional appointment 6 weeks post op and 12 weeks post op, the surgeons have no status of the patient, and no markers to check if the postoperative care is evolving right.

Currently, the investigators are using a mobile application (Orthense by Digikare, Blagnac, France) to complement in-person postoperative follow-up care for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing rotator cuff surgery. They must be able to use a mobile-app, and have an email address and internet connexion.

Exclusion Criteria:

* Unable to read French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Return rate | 6 weeks postoperative
  The overall response rate to the questionnaires

SECONDARY OUTCOMES:
The quality of the responses | 6 weeks postoperative
  response rate inside the questionnaire
Net Promoter Score (NPS) | 6 weeks postoperative
  whether or not the patient recommended the questionnaire used, a scale of 0 (not at all likely) to 10 (very likely)
Overall patient satisfaction | 6 weeks postoperative
  whether or not the patient is satisfied of the questionnaire used, a scale of 0 (not at all) to 10 (very good)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Grimberg, MD, Study Director — L'Institut de Recherche en Chirurgie Orthopédique et Sportive
Locations (1):
- Clinique Jouvenet, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gil JA, Durand WM, Johnson JP, Goodman AD, Owens BD, Daniels AH. Unanticipated Admission Following Outpatient Rotator Cuff Repair: An Analysis of 18,061 Cases. Orthopedics. 2018 May 1;41(3):164-168. doi: 10.3928/01477447-20180501-04. Epub 2018 May 9. PMID 29738599
- [Background] Calvo E, Torres MD, Morcillo D, Leal V. Rotator cuff repair is more painful than other arthroscopic shoulder procedures. Arch Orthop Trauma Surg. 2019 May;139(5):669-674. doi: 10.1007/s00402-018-3100-0. Epub 2018 Dec 17. PMID 30560289
- [Background] Kosinski LR, Gil JA, Durand WM, DeFroda SF, Owens BD, Daniels AH. 30-Day readmission following outpatient rotator cuff repair: an analysis of 18,061 cases. Phys Sportsmed. 2018 Nov;46(4):466-470. doi: 10.1080/00913847.2018.1502571. Epub 2018 Jul 27. PMID 30021075
- [Background] Higgins J, Semple J, Murnaghan L, Sharpe S, Theodoropoulos J. Mobile Web-Based Follow-up for Postoperative ACL Reconstruction: A Single-Center Experience. Orthop J Sports Med. 2017 Dec 22;5(12):2325967117745278. doi: 10.1177/2325967117745278. eCollection 2017 Dec. PMID 29318171
- [Background] Armstrong KA, Coyte PC, Brown M, Beber B, Semple JL. Effect of Home Monitoring via Mobile App on the Number of In-Person Visits Following Ambulatory Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 Jul 1;152(7):622-627. doi: 10.1001/jamasurg.2017.0111. PMID 28329223
- [Derived] Descamps J, Le Hanneur M, Bouche PA, Boukebous B, Duranthon LD, Grimberg J. Do web-based follow-up surveys have a better response rate than traditional paper-based questionnaires following outpatient arthroscopic rotator cuff repair? A randomized controlled trial. Orthop Traumatol Surg Res. 2023 Apr;109(2):103479. doi: 10.1016/j.otsr.2022.103479. Epub 2022 Nov 17. PMID 36403889